CLINICAL TRIAL: NCT02461654
Title: EuroPainClinics® Study III (Prospective Observational Study)
Acronym: EPCSIII
Status: Terminated | Type: Observational
Why Stopped: The clinical trial was suspended for the reason that preliminary results in 20 patients didn't show a significant curative effect of observed treatment.
Sponsor: Europainclinics z.ú. (Other)
Responsible Party: Sponsor
Other Study IDs: 9N-2015
Record Dates: First submitted 2015-05-26; First posted 2015-06-03 (Estimated); Last update posted 2022-01-13 (Actual); Status verified 2021-12

CONDITIONS: Disc Herniations
MeSH Terms: conditions — Intervertebral Disc Displacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Disc FX — Disc FX is an innovative system allowing for a safe and effective approach to a damaged disc without injury to the surrounding structures. The procedure consists of three phases: during the first phase, the disc is punctured with a special needle that functions as a working channel. This needle is used to remove part of the degenerate inner tissue. Then, using a radio-frequency probe, the disc is sealed to minimize the risk of repeated herniation. In the final step, the pathological nerves in the back part of the disc are destroyed with the use of radio-frequency.

SUMMARY:
In this prospective observational trial the effect of the Disc FX microinvasive therapy should be examined in (approximately 150) adult patients with low back pain.

DETAILED DESCRIPTION:
Patients will be selected from 4 participating clinics from Czech and Slovak republic. Trial will compare evolution of patient's health state, changes of low back pain and other neurological conditions during time period (6 and 12 month) after miniivasive interventional pain release procedure - disc FX.

Back pain due to Lumbar Disc Disease in our population is a very common problem. The treatment options range from physiotherapy to fusion surgery. When all conservative treatment is failed than in some cases with suitable conditions of intervertebral disc is possible to avoid classical disc surgery with minimally invasive surgery techniques. A number of minimally invasive procedures have also been developed in the recent past for its management. One of them is Disc FX procedure. Disc FX is an innovative system allowing for a safe and effective approach to a damaged disc without injury to the surrounding structures. This method provides an option for those people who have not benefited from conservative treatment, and are not yet ready for major surgery. It is a minimal-access procedure performed on an out-patient basis. Its big advantage is the fact that the patient may go home the same day. The procedure consists of three phases: during the first phase, the disc is punctured with a special needle that functions as a working channel. This needle is used to remove part of the degenerate inner tissue. Then, using a radio-frequency probe, the disc is sealed to minimize the risk of repeated herniation. In the final step, the pathological nerves in the back part of the disc are destroyed with the use of radio-frequency.

Trial will compare evolution of patient's health state, changes of low back pain and other neurological conditions during time period (6 and 12 month) after miniivasive interventional pain release procedure - disc FX.

ELIGIBILITY:
Inclusion Criteria:

* Patients who undergo Disc FX therapy

Exclusion Criteria:

* No

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Trial will compare evolution of patient's health state, changes of low back pain and other neurological conditions during time period (6 and 12 month) after miniivasive interventional algesiologic procedure - disc FX.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2018-12-31 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Pain as assessed by the Visual analogue scale | 3 years
  All acquired information will be noted in to the special anonymous protocol

SECONDARY OUTCOMES:
Pain localization as assessed by note of radiating dermatome as neurologic examination | 3 years
  All acquired information will be noted in to the special anonymous protocol
Pain progress as assessed by global pain scale | 3 years
  All acquired information will be noted in to the special anonymous protocol
Changes in analgesics drugs consumption as assessed by equianalgesic dose ratios for opioids | 3 years
  All acquired information will be noted in to the special anonymous protocol

CONTACTS AND LOCATIONS:
Overall Officials: Juraj Mláka, MD PhD, Study Chair — R-Clinic; Ladislav Kočan, MD PhD, Study Director — K-medicine
Locations (1):
- Algesiology ambulance, Prague, Czechia